CLINICAL TRIAL: NCT04436315
Title: Intervention Study of an Individualized Exergame Training for People With Major Neurocognitive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Davy Vancampfort (Other)
Responsible Party: Sponsor-Investigator, Davy Vancampfort, Professor, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 082020
Record Dates: First submitted 2020-06-03; First posted 2020-06-18 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Exergame; Major Neurocognitive Disorder; Long-term Care Facility; Nursing Home

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Exergame intervention
  Interventions: Device: Motor-cognitive training device
- Control (Sham Comparator): Active control condition
  Interventions: Other: Active control condition

INTERVENTIONS:
Device: Motor-cognitive training device — Motor-cognitive training device
  Other Names: Vitaal exergame
  Arms: Intervention
Other: Active control condition — Physical activity program
  Other Names: Physical therapy program
  Arms: Control

SUMMARY:
This study evaluates the feasibility of the intervention and the study design.

DETAILED DESCRIPTION:
This study evaluates the feasibility of the intervention and the study design. Furthermore, it investigates the effects of an exergame training including strength, balance, cognitive and pelvic floor muscle training. The main risk in this study is related to potential accidents/falls during the training (and not mainly to the data acquisition procedures). But as the difficulty of the training game is adaptive, the participants will always be challenged on an appropriate level for their physical condition. Furthermore, before and after the training period, several low risk measurements are conducted. This study contributes to fundamental research investigating how multicomponent exergame training influence physical and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60+ years
* Living in residency "de Wingerd" in Leuven (at least two weeks here)
* Being able to straight for minimal 10 minutes without aids
* Visual acuity with correction sufficient to see on a TV screen
* diagnosed with major neurocognitive disorder

Exclusion Criteria:

* Mobility impairments that don't allow to play the exergame
* Any unstable cardiovascular or other health condition which according to the American College of Sports Medicine Standards might lead to unsafe participation (e.g. recent cardiac infarction, uncontrolled diabetes or hypertension)
* Orthopaedic or neurological diseases that prevent exergame training
* Rapidly progressive or terminal illness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 2 years
  Recruitment rate Adherence Attrition Time management of the assessments during pre-/post-measurements and the intervention Safety
Motor functions | 2 years
  Recruitment rate Adherence Attrition Time management of the assessments during pre-/post-measurements and the intervention Safety Short Physical Performance Battery
  1 - Minute Sit to Stand Test
Cognitive functions | 2 years
  Montréal Cognitive Assessment Mini-Mental State Examination
Mental health | 2 years
  Cornell Scale for Depression in Dementia Neuropsychiatric Inventory Dementia Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- De Wingerd, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swinnen N, de Bruin ED, Guimaraes V, Dumoulin C, De Jong J, Akkerman R, Vandenbulcke M, Stubbs B, Vancampfort D. The feasibility of a stepping exergame prototype for older adults with major neurocognitive disorder residing in a long-term care facility: a mixed methods pilot study. Disabil Rehabil. 2023 Feb 23:1-15. doi: 10.1080/09638288.2023.2182916. Online ahead of print. PMID 36824039